CLINICAL TRIAL: NCT06553365
Title: An Open, Single-Arm Phase II Study Evaluating the Efficacy and Safety of FCN-159 in Selected NF2-associated Nerve Sheath Tumors
Brief Title: Phase II Study of FCN-159 in NF2 Nerve Sheath Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-159-IIT02
Record Dates: First submitted 2024-08-03; First posted 2024-08-14 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Nerve Sheath Tumor
Keywords: MEK; NF2; nerve sheath tumor
MeSH Terms: conditions — Nerve Sheath Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCN-159 (Experimental): FCN-159 8mg qd po
  Interventions: Drug: FCN-159

INTERVENTIONS:
Drug: FCN-159 — FCN-159 8mg qd po

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of FCN-159 in patients with specific NF2-associated nerve sheath tumors.

DETAILED DESCRIPTION:
1. A phase 2 single arm single center study, total 30 patients will be enrolled;
2. To evaluate the safety and efficacy of FCN-159, a Mek inhibitor, to treat NF2; associated nerve sheath tumors, age≥16, including benign and malignant tumors;
3. Primary endpoint: Objective response rate (ORR)；Secondary Outcome Measures： Clinical benefit rate (CBR)；24w WRS, OS et al..

ELIGIBILITY:
Inclusion Criteria:

1. ≥16 years of age, regardless of gender.
2. meet the revised 2022 diagnostic criteria for NF2-associated nerve sheath tumors or pathologically confirmed NF2-associated nerve sheath tumors.
3. should meet one of the following criteria: 1) Incomplete surgical resection, or postoperative recurrence. 2) Systemic therapy is required as determined by the Investigator.
4. the presence of a measurable lesion, as defined by REiNS or RECIST V1.1 criteria.
5. Karnofsky physical status score of ≥70.
6. the patient has adequate organ and bone marrow function.
7. International Normalized Ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN.
8. For patients of childbearing potential: During treatment and for at least 90 days after the last dose, patients should agree to use a highly effective method of contraception.
9. avoid excessive sun exposure and be willing to use an adequate amount of sunscreen in anticipation of sun exposure.
10. be able to understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

* Previously received one of the following treatments:

  1. Pharmaceutical or biological therapy within 3 weeks or 5 half-lives prior to enrollment, whichever is longer.
  2. Use of growth factors that promote platelet, red blood cell, or white blood cell count or function within 7 days prior to enrollment.
  3. Patients who have received major surgery or anti-tumor immunotherapy within 4 weeks prior to enrollment.
  4. Radiation therapy for nerve sheath tumors within 4 weeks prior to enrollment.
  5. Dose adjustment for patients treated with dexamethasone or other corticosteroids within 1 week prior to enrollment.
  6. Patients who have participated in another interventional clinical trial within 4 weeks prior to enrollment.
  7. Prior treatment with Selumetinib or any other MEK 1/2 inhibitor. 2. history of or concurrent with other malignancies. 3. inability to undergo MRI and/or contraindications to MRI. 4. uncontrolled hypertension. 5. the presence of dysphagia, active gastrointestinal disease, malabsorption syndrome, or other condition that interferes with the absorption of the study medication.

     6. previous or current retinal vascular disease. 7. interstitial pneumonitis 8. cardiac function or co-morbidities 9. Immediate family history of sudden cardiac death before age 50. 10.History of any acute neurological condition 11. with active bacterial, fungal or viral infections 12. known hypersensitivity to the study drug, other MEK1/2 inhibitors, or their excipients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) estimated by investigators | Every 4 cycles (each cycle is 28 days), assessed up to 2 years
  Investigator-assessed objective mitigation rate ORR (Reponse evaluation in Nerufibromatosis and Schwannomatosis, REiNS criteria and RECIST 1.1 criteria, respectively)

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) estimated by investigators | Every 4 cycles (each cycle is 28 days), assessed up to 2 years
  Clinical benefit rate CBR will be assessed by the investigator (REiNS criteria and RECIST 1.1 criteria respectively)
24-week word recognition score (WRS) | up to 24 weeks
  Hearing response changes will be assessed in patients with hearing impairment (24-week word recognition scores and pure tone audiometry).
pain estimated by NRS | Every 4 cycles (each cycle is 28 days), assessed up to 2 years
  Change in pain intensity score relative to baseline will be assessed according to NRS scale.
Duration of response (DOR) assessed by investigator | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Duration of response (DoR) is estimated by the investigators as the time from treatment initiation to disease progression or death in patients who achieve complete or partial response, using both RECIST V1.1 and REINS criteria.
progression free survival (PFS) assessed by investigator | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  PFS is estimated by the investigators as the time from treatment initiation to disease progression or death in patients, using both RECIST V1.1 and REINS criteria.

OTHER OUTCOMES:
life quality assessed by NFTI-QOL | Every 4 cycles (each cycle is 28 days), assessed up to 2 years
  Change in quality of life scores relative to baseline will be assessed by Neurofibromatosis type 2 impact on quality of life (NFTI-QOL) score. The higher score means worse life quality.
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE 5.0 | During the intervention
  Adverse events during treatment of FCN-159 will be assessed by the investigators accroding to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang wang, PhD, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Shuhang Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
the decision will be made after the primary analysis of results.